CLINICAL TRIAL: NCT01572207
Title: Using Targeted Print-material to Promote Physical Activity Behavior in Adults With Multiple Sclerosis
Brief Title: Promoting Physical Activity Behavior in Persons With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Matthew Plow, Project Scientist, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10-531; 1R03HD060073-01A1 (NIH)
Record Dates: First submitted 2012-03-28; First posted 2012-04-06 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Exercise; Physical activity; Quality of life
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate Exercise (Experimental): Subjects assigned to the immediate group will be prescribed a home exercise program during the first meeting. During the 12 week training period, the subject will read pamphlets (sent by mail) once to twice a month about developing skills to manage MS symptoms and motivational pamphlets about physical activity. In addition, the subject will have a phone conversation every two to three weeks with research staff to discuss the progress of the exercise program and to complete a short survey about his/her physical activity level.
  Interventions: Behavioral: Immediate exercise
- Delayed exercise (Experimental): Subjects assigned to the delayed group will be asked to begin the same home exercise program 12 weeks following the first meeting. During the 12 week training period, the subject will receive pamphlets, have phone conversations with research staff, and complete physical activity surveys as described above.
  Interventions: Behavioral: Delayed exercise

INTERVENTIONS:
Behavioral: Immediate exercise — Subjects in the immediate exercise group will be prescribed a home exercise program during the first meeting and will begin the 12 week training period immediately following the first meeting.
  Other Names: Treatment arm
  Arms: Immediate Exercise
Behavioral: Delayed exercise — Subjects in the delayed exercise group will begin the home exercise program 12 weeks following the initial meeting.
  Other Names: control arm
  Arms: Delayed exercise

SUMMARY:
The purpose of this research study is to evaluate whether tailored print material can promote physical activity and exercise, and subsequently improve quality of life and fitness levels among people with multiple sclerosis (MS). Research suggests that routine physical activity is beneficial in people with mild to moderate MS. However, people with MS may face many barriers for engaging in regular physical activity. Prescribing a home exercise program and receiving tailored motivational print material may help people engage in physical activity. Thus, the investigators hope to figure out whether tailored print material can be used as strategy to promote physical activity and improve physical function in people with MS.

DETAILED DESCRIPTION:
The objective of the proposed study is to further our understanding of methods to promote physical activity (PA) in people with multiple sclerosis (MS). The investigators will evaluate the efficacy of a print-based multifaceted intervention that consists of prescribing an exercise program and teaching self-management strategies.

ELIGIBILITY:
Inclusion Criteria:

* A physician-confirmed diagnosis of relapsing-remitting MS

Exclusion Criteria:

* Exercise more than 150 minutes per week
* Pregnant
* Metabolic or cardiopulmonary disease that puts patient at high risk for engaging in a home exercise program (patients with controlled diabetes and high blood pressure will still be considered eligible)
* Four or more falls in the past 6 months
* Be able to walk 25 feet with or without a cane
* Severe cognitive deficits
* Unable to read at a 6th grade level
* A condition besides MS that had lead to hospitalization in the past year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Plow, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- The Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Immediate Exercise | Delayed Exercise
Started | 14 | 16
Completed | 12 | 13
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Exercise | Delayed Exercise | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 16 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (9) | 48 (10) | 47.5 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 16 | 30

OUTCOME MEASURES:

1. Primary Outcome: Changes From Baseline in Physical Activity Behavior
Description: Physical activity behavior will be measured with the Godin Leisure-Time Exercise Questionnaire. The Godin Leisure-Time Exercise Questionnaire calculates total weekly leisure activity by summing the products of separate intensities. Weekly leisure activity score = (9 x time/week) + (5 x times/week) + (3 x times/week) for strenuous, moderate and light activities, respectively. The scale is summed to equal the Total Units Mean.
  With this scale, higher numbers are considered to be the better outcome as it indicates more physical activity.
Time Frame: Each subject will be given the questionnaire at 3 points during the study, at baseline, interim test (an average of 12 weeks from baseline) and at posttest (an average of 24 weeks from baseline).
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | Immediate Exercise | Delayed Exercise
Number analyzed (Participants) | 14 | 16
scores on a scale
  Total Score (Week 1 - baseline) | 14.36 [0 to 36] | 16.22 [0 to 64]
  Total Score (Week12) | 33.07 [0 to 85] | 21.00 [0 to 45]
  Total Score (Week 24) | 26 [0 to 58] | 23.06 [3 to 43]

2. Secondary Outcome: Changes From Baseline in Physical Fitness
Description: The physical assessment will include measuring the 6-minute walk test. The units reported are in meters for distance traveled by each participant during the six minutes. For this scale, the higher number is the better score as it is a direct measure of distance traveled.
Time Frame: Each patient will be given the assessment at 3 points during the study, at baseline, interim test (an average of 12 weeks from baseline) and at posttest (an average of 24 weeks from baseline).
Measure: Mean (Full Range); unit: meters
Arm/Group | Immediate Exercise | Delayed Exercise
Number analyzed (Participants) | 14 | 16
meters
  6-minute walk (Week 1 - baseline) | 382.56 [213.36 to 489.66] | 324.12 [144.17 to 483.72]
  6-minute walk (Week 12) | 407.03 [207.90 to 507.64] | 321.23 [91.44 to 464.82]
  6-minute walk (Week 24) | 406.42 [207.90 to 558.55] | 333.09 [139.02 to 479.15]

3. Secondary Outcome: Changes From Baseline in Quality of Life
Description: The Multiple Sclerosis Impact Scale will be administered. The total score is a sum of individual question scores, ranging from 29 (best possible outcome) to 145 (worst possible outcome). Therefore, the lower the number, the better the outcome.
Time Frame: as for outcome 2
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | Immediate Exercise | Delayed Exercise
Number analyzed (Participants) | 14 | 16
scores on a scale
  MS Impact score (Week 1 - baseline) | 58.57 [31 to 98] | 62.31 [30 to 106]
  MS Impact score (Week 12) | 53.57 [30 to 85] | 67.13 [33 to 119]
  MS Impact score (Week 24) | 52.29 [29 to 114] | 65.38 [31 to 122]

ADVERSE EVENTS:
Arm/Group | Immediate Exercise | Delayed Exercise
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/16
Other Adverse Events (participants affected / at risk) | 0/14 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No